CLINICAL TRIAL: NCT04793919
Title: Treatment Study for Children and Adolescents With Acute Promyelocytic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Associazione Italiana Ematologia Oncologia Pediatrica (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICC APL STUDY 02; 2017-002383-40 (EudraCT Number)
Record Dates: First submitted 2019-11-13; First posted 2021-03-11 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Acute Promyelocytic Leukemia
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Gemtuzumab; Arsenic Trioxide; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Risk (SR) (Active Comparator): Patient with APL and WBC less than 10x10e9/L at presentation before start treatment
  Interventions: Drug: Arsenic Trioxide; Drug: All-trans retinoic acid
- High Risk (HR) (Experimental): Patient with APL, with the highest pre-treatment WBC count equal to or greater than 10x10e9/L at presentation
  Interventions: Drug: Mylotarg; Drug: Arsenic Trioxide; Drug: All-trans retinoic acid

INTERVENTIONS:
Drug: Mylotarg — See the protocol
  Other Names: GO
  Arms: High Risk (HR)
Drug: Arsenic Trioxide — See the protocol
  Other Names: ATO
Drug: All-trans retinoic acid — See the protocol
  Other Names: ATRA

SUMMARY:
The trial is open to all patients with a diagnosis of acute promyelocytic leukemia (APL) who are PCR-positive for the PML-RARα transcript and less than 18 years of age.

DETAILED DESCRIPTION:
Acute promyelocytic leukemia (APL) in children has become a highly curable disease with the combination of all-trans retinoic acid (ATRA) and anthracycline-based chemotherapy with an overall remission rates equal to or higher than 98% and cure rates now exceeding 80% 1-9.

Based on data coming from adults indicating that at least standard-risk APL patients may be cured without chemotherapy (i.e., with a treatment combining arsenic trioxide (ATO) and ATRA only) 10-12, this ICC APL 02 study was designed with the aim of validating the efficacy of a treatment combining:

* ATO and ATRA in newly diagnosed APL standard-risk (SR) children and adolescents and
* ATO, ATRA and gemtuzumab ozogamicin (GO) in newly diagnosed APL high-risk (HR) children and adolescents.

Following one induction course of treatment combining ATO and ATRA +/- GO depending on risk stratification, patients will receive 4 ATO/ATRA based consolidation blocks. This is the first pediatric trial delivering a non-chemotherapy-based treatment for children with APL, being the whole treatment based on the use of ATRA, ATO (and GO in HR patients). The aim of the study is to demonstrate at least an equivalent efficacy and safety of this treatment not containing cytostatic agents compared to the standard protocols combining ATRA and chemotherapy (i.e. ICC APL Study 01).

The trial is open to all patients with a diagnosis of acute promyelocytic leukemia (APL) who are PCR-positive for the PML-RARα transcript and less than 18 years of age.

This will be an international study, comprising the most important pediatric European groups, expecting to recruit 46 and 43 patients in SR and HR arms, respectively, in 3 years. The duration of study recruitment will be 36 months with a minimum follow-up per patient of 2 years.

The evaluation of morphological CR will be carried out after induction therapy, prior to the first block of consolidation therapy. MRD results after induction will not have an impact on subsequent therapy. By contrast, MRD results after the third consolidation course will influence the subsequent treatment, MRD-positive patients being eligible to rescue treatment, including hematopoietic stem cell transplantation (HSCT). BM aspirates will be repeated after the end of therapy, and 3 months, 6 months, 9 months and 12 months after treatment discontinuation.

This is a collaborative international study in APL in children and adolescents aimed at providing information about procedures for the entry, treatment and follow-up of pediatric patients with APL. It is not intended that this document be used as an aide-memoir or guide for the treatment of other patients. Every care has been taken in its drafting, but corrections and amendments may be necessary. Before entering patients into the study, clinicians must ensure that the study has received clearance from their Local Research Ethics Committee and any other necessary body.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed APL confirmed by the presence of PML/RARα fusion gene
* Age <18 years
* Written informed consent by parents or legal guardians

Exclusion Criteria:

* Patients with a clinical diagnosis of APL but subsequently found to lack PML/RARα rearrangement should be withdrawn from the study and treated on an alternative protocol
* Significant liver dysfunction (bilirubin serum levels >3 mg/dL, ALT/AST serum levels greater than 5 times the normal values)
* Creatinine serum levels >2 times the normal value for age
* Significant arrhythmias, EKG abnormalities (*see below), other cardiac contraindications (L-FEV <50% or LV-FS <28%)
* Neuropathy
* Concurrent active malignancy
* Uncontrolled life-threatening infections
* Pregnant or lactating female
* Patients who had received alternative therapy (APL not initially suspected; ATRA and/or ATO not available

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 89 (Estimated)
Dates: Start 2019-10-09 (Actual); Primary Completion 2025-10-09 (Estimated); Study Completion 2027-10-10 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival (EFS) probability | 3 years
  SR patients: To evaluate the efficacy in terms of event-free survival of a treatment combining arsenic trioxide (ATO) and all-trans retinoic acid (ATRA) in newly diagnosed APL standard-risk children and adolescents HR patients: To evaluate the efficacy in terms of event-free survival of a treatment combining arsenic trioxide (ATO), all-trans retinoic acid (ATRA) and gemtuzumab ozogamicin (GO) in newly diagnosed APL high-risk children and adolescents

SECONDARY OUTCOMES:
Rate of hematological CR/CRi after induction | 5 years
  To evaluate the rate of hematological Complete Remission (CR) (defined as bone marrow regenerating normal hematopoietic cells and containing < 5% blast cells by morphology, with ANC in peripheral blood > 1.0 x 10^9/L and platelet count > 100 x 10^9/L) and Complete Remission with incomplete hematologic recovery (CRi) (defined as CR except that peripheral blood neutrophils and/or platelets do not meet the criteria as defined above) after induction therapy.
Rate of molecular CR/CRi after induction | 5 years
  To evaluate the rate of molecular CR/CRi (defined as the absence of PML/RARα fusion transcript in bone marrow assessed by RQ-PCR, with an assay sensitivity of at least 10^-4).
Rate of early death during induction | 5 years
  To evaluate the rate of early death during induction (defined as any death occurring within 14 days from diagnosis from any cause).
Probability of overall survival (OS) at 3 years | 3 years
  To evaluate the rate of overall survival
Cumulative incidence of relapse (CIR) at 3 years | 3 years
  To evaluate the cumulative incidence of hematological relapse (defined as reappearance of promyeloblasts/abnormal promyelocytes > 5% in the bone marrow) and molecular relapse (defined as reappearance of PML/RARα fusion transcript in two successive samples taken at least 2 weeks apart in patients previously in molecular remission).
Incidence of hematological and non-hematological toxicity | 5 years
  Incidence of treatment-related hematological and non-hematological toxicity assessed by CTCAE v4.0
Rate of molecular remission after 3 consolidation cycles | 5 years
  To evaluate the rate of molecular remission (defined as the absence of PML/RARα fusion transcript in bone marrow assessed by RQ-PCR, with an assay sensitivity of at least 10^-4) after 3 consolidation cycles.
Assessment of PML/RARα transcription level reduction during treatment | 5 years
  To evaluate the reduction of PML/RARα fusion transcript in bone marrow by means of RQ-PCR during treatment.
Pediatric Quality of Life assessment | 5 years
  Pediatric Quality of life assessed by PedsQoL questionnaire, in the questionnaire there is a list of things that might be a problem for the child. The minimum value is 0 (never a problem) - maximum value 4 (almost always problem)
Total hospitalization days during therapy | 5 years
  Number of total hospitalization days during the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Fanco Locatelli, Prof, Principal Investigator — Dept. of Pediatric Hematology Oncology - Bambino Gesù Children's Hospital Rome
Locations (31):
- Hôpital Universitaire des Enfants Reine Fabiola (Huderf), Brussels, Belgium
- University Hospital Motol, Prague, Czechia
- Pediatrics and Adolescent Medicine Aarhus University Hospital, Aarhus N, Denmark
- CHU de Bordeaux - Hôpital des Enfants, Bordeaux, France
- Universitätsklinikum Essen (AöR) Zentrum für Kinder-und Jugendmedizin Klinik für Kinderheilkunde III, Essen, Germany
- Our Lady's Children's Hospital Crumlin, Dublin, Ireland
- Rappaport Children'S Hospital, Rambam Health Care Campus, Haifa, Israel
- Italy (18):
  - Ospedale "Casa Sollievo della Sofferenza" - UO Oncoematologia Pediatrica, San Giovanni Rotondo, Foggia
  - AOU Policlinico Dipartimento di Pediatria, Bari
  - Ospedale Papa Giovanni XXIII - USS Oncoematologia Pediatrica, Bergamo
  - AOU Policlinico Sant'Orsola-Malpighi - Oncologia ed Ematologia Pediatrica, Bologna
  - Ospedale Pediatrico Microcitemico "A.Cau", Az.Ospedaliera Brotzu - SC Oncoematologia Ped. e Patologia della coagulazione, Cagliari
  - AOU Policlinico Vittorio Emanuele - UOC Ematologia ed Oncologia Pediatrica con TNO, Catania
  - A.O. Universitaria Meyer - DAI Oncoematologia Pediatrica, Florence
  - IRCCS Istituto Gannina Gaslini - Dipartimento di Oncoematologia, Genova
  - Fondazione Monza e Brianza per il Bambino e la sua Mamma (MBBM) - Ospedale San Gerardo, Monza
  - AORN Santobono-Pausilipon, Napoli
  - Univerità degli Studi della Campania- Luigi Vanvitelli - Sevizio di Oncologia Pediatrica, Napoli
  - Azienda Ospedaliera di Padova - Oncoematologia Pediatrica, Padua
  - ARNAS Civico di Cristina e Benfratelli - UOC Oncoematologia Pediatrica, Palermo
  - Fondazione IRCCS Policlinico San Matteo - Oncoematologia Pediatrica, Pavia
  - Ospedale santa Chiara - AOU Pisana, UO Oncoematologia Pediatrica, Pisa
  - Policlinico Umberto I Università "LA Sapienza" - Dip. Biotecnologie cellulari ed ematologia UOS Ematologia Pediatrica, Roma
  - Dipartimento di Onco-Ematologia e Terapia Cellulare e Genica - Ospedale Pediatrico "Bambino Gesù", Roma
  - AOU Città della Salute e della Scienza di Torino - Presidio Infantile Regina Margherita, Torino
- VU medisch centrum, Amsterdam, Netherlands
- Portugal (3):
  - Centro Hospitalar Universitário de Coimbra - Hospital Pediátrico de Coimbra, Coimbra
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, EPE, Lisbon
  - Instituto Português de Oncologia do Porto Francisco Gentil, E. P. E., Porto
- Valencia University Medical School University Hospital La Fe, Valencia, Spain
- Childrens hematology and oncology Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No